CLINICAL TRIAL: NCT02387359
Title: A Randomized, 12-Week, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Plecanatide in Patients With Irritable Bowel Syndrome With Constipation (IBS-C)
Brief Title: The Plecanatide Irritable Bowel Syndrome With Constipation Study (IBS-C)
Acronym: IBS-C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP304203-04
Record Dates: First submitted 2015-01-20; First posted 2015-03-13 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Irritable Bowel Syndrome Characterized by Constipation
MeSH Terms: interventions — plecanatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3.0 mg plecanatide (Active Comparator): Plecanatide 3.0 mg dosed daily for 12 weeks
  Interventions: Drug: Plecanatide
- 6.0 mg plecanatide (Active Comparator): Plecanatide 6.0 mg dosed daily for 12 weeks
  Interventions: Drug: Plecanatide
- Matching placebo (Active Comparator): Placebo dosed daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Plecanatide
  Arms: 3.0 mg plecanatide; 6.0 mg plecanatide
Drug: Placebo
  Arms: Matching placebo

SUMMARY:
This study in patients with IBS-C is a randomized, double-blind, placebo-controlled, parallel-group clinical trial with 12 weeks of study drug therapy.

DETAILED DESCRIPTION:
This study in patients with IBS-C is a randomized, double-blind, placebo-controlled, parallel-group clinical trial with 12 weeks of study drug therapy.

Screening/Baseline: Patients will undergo an up to 28-day Screening/Baseline period to allow for any necessary diagnostic procedures, allow for required washout of medications and to determine study eligibility. If otherwise eligible based on screening criteria, patients will undergo a 2-week baseline assessment using an electronic diary where they will record daily assessments of bowel movements (BMs), stool consistency (Bristol Stool Form Scale-BSFS), abdominal pain and other IBS-related symptoms. Data from the two-week electronic diary assessment just prior to the randomization visit will be used to confirm IBS-C and study eligibility as well as define the patient's baseline from which change will be determined.

Treatment: Patients who meet all entry criteria will be randomized (1:1:1) to one of three blinded treatment groups on Day 1 of the Treatment period. Patients will take an oral dose of study drug OD for 12 weeks and continue the daily electronic diaries (BMs, rescue medication use, abdominal pain, and other symptoms). During treatment weeks 4, 8, and 12, patients will return to the clinic to undergo safety and efficacy assessments.

Post-Treatment: For 2 weeks after completing dosing, patients will continue to complete daily electronic diaries. Patients will then return to the clinical site for a final follow-up visit during Week 14 following randomization.

The planned duration of participation in this study will be at least 116 days from signing of informed consent through post-treatment or up to approximately 135 days with visit windows considered.

ELIGIBILITY:
Inclusion Criteria:

•Adult patients between the ages of 18 and 85 years (inclusive) with a diagnosis of IBS based on ROME III diagnostic criteria and meeting criteria for diagnosis of the constipation predominant subtype - IBS-C

Exclusion Criteria:

* Refusal or inability to sign informed consent for the trial
* Refusal or inability to complete daily Episodic (real-time) BM / RM calls, End of Day daily Calls, and/or complete electronic questionnaires
* BMI > 35 or < 18
* Women of child bearing potential who refuse to use an acceptable method of birth control for the duration of the trial
* Women who are pregnant or lactating
* Diagnosis of IBS-D or IBS-M
* Organic or obstructive disease of the small or large intestine
* Use of laxatives other than the study-supplied rescue medication (Dulcolax®, bisacodyl)
* Use of a prohibited concomitant medication within the time frame prior to screening outlined in the study protocol for that medication
* Unstable medical illness
* Bilirubin > 3X ULN in the absence of a conjugation defect
* Any laboratory value > 3X ULN unless discussed and approved by the study Medical Monitor

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1054 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul F.C. Eng, PhD, Study Director — Synergy Pharmaceuticals Inc.
Locations (145):
- United States (145):
  - Synergy Research Site, Athens, Alabama
  - Synergy Research Site, Birmingham, Alabama
  - Synergy Research Site, Dothan, Alabama
  - Synergy Research Site, Foley, Alabama
  - Synergy Research Site, Huntsville, Alabama
  - Synergy Research Site, Montgomery, Alabama
  - Synergy Research Site, Chandler, Arizona
  - Synergy Research Site, Glendale, Arizona
  - Synergy Research Site, Phoenix, Arizona
  - Synergy Research Site, Tucson, Arizona
  - Synergy Research Site, Conway, Arkansas
  - Synergy Research Site, Little Rock, Arkansas
  - Synergy Research Site, Anaheim, California
  - Synergy Research Site, Artesia, California
  - Synergy Research Site, Chula Vista, California
  - Synergy Research Site, Corona, California
  - Synergy Research Site, Encino, California
  - Synergy Research Site, Fountain Valley, California
  - Synergy Research Site, Fresno, California
  - Synergy Research Site, Garden Grove, California
  - Synergy Research Site, La Mesa, California
  - Synergy Research Site, La Mirada, California
  - Synergy Research Site, Laguna Hills, California
  - Synergy Research Site, Lancaster, California
  - Synergy Research Site, North Hollywood, California
  - Synergy Research Site, Sacramento, California
  - Synergy Research Site, San Bernardino, California
  - Synergy Research Site, San Diego, California
  - Synergy Research Site, Thousand Oaks, California
  - Synergy Research Site, Upland, California
  - Synergy Research Site, Broomfield, Colorado
  - Synergy Research Site., Centennial, Colorado
  - Synergy Research Site, Bristol, Connecticut
  - Synergy Research Site, Hamden, Connecticut
  - Synergy Research Site, Boynton Beach, Florida
  - Synergy Research Site, Brandon, Florida
  - Synergy Research Site, DeLand, Florida
  - Synergy Research Site, Fort Lauderdale, Florida
  - Synergy Research Site, Homestead, Florida
  - Synergy Research Site, Inverness, Florida
  - Synergy Research Site, Jacksonville, Florida
  - Synergy Research Site, Miami, Florida
  - Synergy Research Site, Miami Lakes, Florida
  - Synergy Research Site, Miami Springs, Florida
  - Synergy Research Site, Orlando, Florida
  - Synergy Research Site, Ormond Beach, Florida
  - Synergy Research Site, Oviedo, Florida
  - Synergy Research Site, Port Orange, Florida
  - Synergy Research Site, St. Petersburg, Florida
  - Synergy Research Site, Tampa, Florida
  - Synergy Research Site, Atlanta, Georgia
  - Synergy Research Site, Marietta, Georgia
  - Synergy Research Site, Norcross, Georgia
  - Synergy Research Site, Stockbridge, Georgia
  - Synergy Research Site, Idaho Falls, Idaho
  - Synergy Research Site, Chicago, Illinois
  - Synergy Research Site, Evanston, Illinois
  - Synergy Research Site, Evergreen Park, Illinois
  - Synergy Research Site, Rockford, Illinois
  - Synergy Research Site, Evansville, Indiana
  - Synergy Research Site, Augusta, Kansas
  - Synergy Research Site, Newton, Kansas
  - Synergy Research Site, Topeka, Kansas
  - Synergy Research Site, Wichita, Kansas
  - Synergy Research Site, Baton Rouge, Louisiana
  - Synergy Research Site, Crowley, Louisiana
  - Synergy Research Site, Mandeville, Louisiana
  - Synergy Research Site, Metairie, Louisiana
  - Synergy Research Site, Monroe, Louisiana
  - Synergy Research Site, New Orleans, Louisiana
  - Synergy Research Site, Shreveport, Louisiana
  - Synergy Research Site, Baltimore, Maryland
  - Synergy Research Site, Hagerstown, Maryland
  - Synergy Research Site, Boston, Massachusetts
  - Synergy Research Site, Chesterfield, Michigan
  - Synergy Research Site, Flint, Michigan
  - Synergy Research Site, Rochester, Michigan
  - Synergy Research Site, Wyoming, Michigan
  - Synergy Research Site., Jackson, Mississippi
  - Synergy Research Site, Hazelwood, Missouri
  - Synergy Research Site, Omaha, Nebraska
  - Synergy Research Site, Las Vegas, Nevada
  - Synergy Research Site, Marlton, New Jersey
  - Synergy Research Site, Albuquerque, New Mexico
  - Synergy Research Site, Brooklyn, New York
  - Synergy Research Site, Great Neck, New York
  - Synergy Research Site, New Windsor, New York
  - Synergy Research Site, New York, New York
  - Synergy Research Site, North Massapequa, New York
  - Synergy Research Site, Asheboro, North Carolina
  - Synergy Research Site, Cary, North Carolina
  - Synergy Research Site, Charlotte, North Carolina
  - Synergy Research Site, Concord, North Carolina
  - Synergy Research Site, Davidson, North Carolina
  - Synergy Research Site, Greensboro, North Carolina
  - Synergy Research Site, Kinston, North Carolina
  - Synergy Research Site, Lenoir, North Carolina
  - Synergy Research Site, Raleigh, North Carolina
  - Synergy Research Site, Wilmington, North Carolina
  - Synergy Research Site, Winston-Salem, North Carolina
  - Synergy Research Site, Fargo, North Dakota
  - Synergy Research Site, Beavercreek, Ohio
  - Synergy Research Site, Cincinnati, Ohio
  - Synergy Research Site, Cleveland, Ohio
  - Synergy Research Site, Englewood, Ohio
  - Synergy Research Site, Sylvania, Ohio
  - Synergy Research Site, Oklahoma City, Oklahoma
  - Synergy Research Site, Tulsa, Oklahoma
  - Synergy Research Site, Portland, Oregon
  - Synergy Research Site, Levittown, Pennsylvania
  - Synergy Research Site, Philadelphia, Pennsylvania
  - Synergy Research Site, Pittsburgh, Pennsylvania
  - Synergy Research Site, Smithfield, Pennsylvania
  - Synergy Research Site, Uniontown, Pennsylvania
  - Synergy Research Site, Columbia, South Carolina
  - Synergy Research Site, Gaffney, South Carolina
  - Synergy Research Site., Greer, South Carolina
  - Synergy Research Site, North Charleston, South Carolina
  - Synergy Research Site, Rapid City, South Dakota
  - Synergy Research Site, Athens, Tennessee
  - Synergy Research Site, Chattanooga, Tennessee
  - Synergy Research Site, Memphis, Tennessee
  - Synergy Research Site., Nashville, Tennessee
  - Synergy Research Site, Arlington, Texas
  - Synergy Research Site, Austin, Texas
  - Synergy Research Site, Carrollton, Texas
  - Synergy Research Site, Dallas, Texas
  - Synergy Research Site, Houston, Texas
  - Synergy Research Site, Plano, Texas
  - Synergy Research Site, San Antonio, Texas
  - Synergy Research Site, Webster, Texas
  - Synergy Research Site, Bountiful, Utah
  - Synergy Research Site, Ogden, Utah
  - Synergy Research Site, Sandy City, Utah
  - Synergy Research Site, St. George, Utah
  - Synergy Research Site, Alexandria, Virginia
  - Synergy Research Site, Charlottesville, Virginia
  - Synergy Research Site, Lynchburg, Virginia
  - Synergy Research Site, Newport News, Virginia
  - Synergy Research Site, Bellevue, Washington
  - Synergy Research Site, Spokane, Washington
  - Synergy Research Site, Charleston, West Virginia
  - Synergy Research Site, Morgantown, West Virginia
  - Synergy Research Site, Milwaukee, Wisconsin
  - Synergy Research Site, Wauwatosa, Wisconsin

REFERENCES:
- [Derived] Brenner DM, Shin AS, Laitman AP, Deutsch JK, Kunkel DC. The Effectiveness of Plecanatide for Treating Constipation and Bloating in Patients Aged 18 to 40 Years With Irritable Bowel Syndrome: Utilization of a New Composite Trisymptom Endpoint. J Gastroenterol Hepatol. 2025 Dec;40(12):2890-2897. doi: 10.1111/jgh.70119. Epub 2025 Nov 10. PMID 41214272
- [Derived] Cash BD, Sharma A, Walker A, Laitman AP, Chang L. Plecanatide for the treatment of chronic idiopathic constipation and irritable bowel syndrome with constipation: Post hoc analyses of placebo-controlled trials in adults with severe constipation. Neurogastroenterol Motil. 2023 Sep;35(9):e14632. doi: 10.1111/nmo.14632. Epub 2023 Jun 18. PMID 37332239
- [Derived] Menees SB, Franklin H, Chey WD. Evaluation of Plecanatide for the Treatment of Chronic Idiopathic Constipation and Irritable Bowel Syndrome With Constipation in Patients 65 Years or Older. Clin Ther. 2020 Jul;42(7):1406-1414.e4. doi: 10.1016/j.clinthera.2020.05.012. Epub 2020 Jul 10. PMID 32660770

RESULTS

PARTICIPANT FLOW:
Groups:
- Matching Placebo: Placebo tablets dosed once daily for 12 weeks
- 3.0 mg Plecanatide: Plecanatide 3.0 mg tablets dosed once daily for 12 weeks
- 6.0 mg Plecanatide: Plecanatide 6.0 mg tablets dosed once daily for 12 weeks
Period: Overall Study
Arm/Group | Matching Placebo | 3.0 mg Plecanatide | 6.0 mg Plecanatide
Started | 354 | 351 | 349
Completed | 295 | 309 | 293
Not Completed | 59 | 42 | 56

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Matching Placebo | 3.0 mg Plecanatide | 6.0 mg Plecanatide | Total
Number analyzed (Participants) | 354 | 351 | 349 | 1054
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (13.71) | 43.0 (13.76) | 43.2 (13.34) | 43.1 (13.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272 | 267 | 266 | 805
  Male | 82 | 84 | 83 | 249

OUTCOME MEASURES:

1. Primary Outcome: Number of Overall Responders - ITT Population
Description: An Overall Responder was a patient who was a Weekly Responder (i.e., decrease of 30% from baseline for abdominal pain intensity and an increase of at least one complete spontaneous bowel movement in the same week) for at least 6 of the 12 treatment weeks.
Time Frame: 12 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Matching Placebo | 3.0 mg Plecanatide | 6.0 mg Plecanatide
Number analyzed (Participants) | 354 | 351 | 349
Participants | 63 | 106 | 103

2. Primary Outcome: Number of Abdominal Pain Responders for at Least 6 of 12 Treatment Weeks
Description: An Abdominal Pain Intensity Responder was a patient who had a decrease of 30% from baseline for abdominal pain intensity. Baseline was the mean of non-missing abdominal pain scores recorded during the 2-week baseline diary assessment period prior to the first dose of study drug.
Time Frame: 12 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Matching Placebo | 3.0 mg Plecanatide | 6.0 mg Plecanatide
Number analyzed (Participants) | 354 | 351 | 349
Participants | 112 | 145 | 156

3. Primary Outcome: Number of Stool Frequency Responder for at Least 6 of the 12 Treatment Weeks
Description: A Stool Frequency Responder is defined as a patient who experienced an increase of at least one CSBM (complete spontaneous bowel movement) per week from baseline. Baseline was the mean number of CSBMs recorded during the 2-week baseline diary assessment period prior to the first dose of study drug.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Matching Placebo | 3.0 mg Plecanatide | 6.0 mg Plecanatide
Number analyzed (Participants) | 354 | 351 | 349
Participants | 124 | 169 | 157

4. Secondary Outcome: Number of Sustained Efficacy Responders
Description: A Sustained Efficacy Responder was a patient who was an Overall Responder who also was a Weekly Responder, i.e., decreased of 30% from baseline for abdominal pain intensity and increased of at least one CSBM (complete spontaneous bowel movement) in the same week for at least 2 of the 4 weeks in month 3 of the Treatment Period.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Matching Placebo | 3.0 mg Plecanatide | 6.0 mg Plecanatide
Number analyzed (Participants) | 354 | 351 | 349
Participants | 61 | 99 | 96

5. Secondary Outcome: Change From Baseline in Stool Consistency
Description: Change from baseline in stool consistency based upon the Bristol Stool Form Scale (BSFS) Rating 1 to 7. Baseline was the mean BSFS score recorded during the 2-week baseline diary assessment period prior to the first dose of study drug. BSFS Rating 1 to 7:
  1. Separate hard lumps, like nuts (hard to pass)
  2. Sausage-shaped but lumpy
  3. Like a sausage but with cracks on its surface
  4. Like a sausage or snake, smooth and soft
  5. Soft blobs with clear-cut edges (passed easily)
  6. Fluffy pieces with ragged edges, a mushy stool
  7. Watery, no solid pieces, entirely liquid
Time Frame: Baseline and 12-Week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Matching Placebo | 3.0 mg Plecanatide | 6.0 mg Plecanatide
Number analyzed (Participants) | 354 | 351 | 349
score on a scale
  Baseline | 2.06 (1.012) | 2.02 (0.918) | 1.98 (0.913)
  Week 12 change from baseline | 1.06 (1.357) | 1.59 (1.592) | 1.86 (1.593)

6. Secondary Outcome: Change From Baseline in Straining
Description: Change from baseline in Straining Score over the 12-week treatment period. Baseline was the mean of non-missing straining scores recorded during the 2-week baseline diary assessment period prior to the first dose of study drug. The severity of straining during a bowel movement was measured using an 11-point scale (0-10 rating; 0 = no straining; 10 = worst straining).
Time Frame: Baseline and 12-week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Matching Placebo | 3.0 mg Plecanatide | 6.0 mg Plecanatide
Number analyzed (Participants) | 354 | 351 | 349
score on a scale
  Baseline | 6.39 (1.991) | 6.47 (1.828) | 6.50 (1.822)
  Week 12 change from baseline | -1.87 (2.464) | -2.69 (2.422) | -2.88 (2.464)

7. Secondary Outcome: Change From Baseline in CSBM Frequency Rate
Description: Change from baseline over the 12-week Treatment Period in CSBM (Complete Spontaneous Bowel Movement) Frequency Rate (CSBMs/Week). Baseline was the mean number of CSBMs recorded during the 2-week baseline diary assessment period prior to the first dose of study drug.
Time Frame: Baseline and 12-Week
Measure: Mean (Standard Deviation); unit: CSBMs per week
Arm/Group | Matching Placebo | 3.0 mg Plecanatide | 6.0 mg Plecanatide
Number analyzed (Participants) | 354 | 351 | 349
CSBMs per week
  Baseline | 0.23 (0.440) | 0.22 (0.465) | 0.28 (0.527)
  Week 12 change from baseline | 0.86 (1.904) | 1.46 (2.565) | 1.41 (2.586)

8. Secondary Outcome: Number of Patients With a SBM Within 24 Hours After the First Dose
Description: Number of patients with a SBM (spontaneous bowel movement) within 24 hours after the first dose of study drug
Time Frame: Up to 24 hours after first dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Matching Placebo | 3.0 mg Plecanatide | 6.0 mg Plecanatide
Number analyzed (Participants) | 354 | 351 | 349
Participants | 118 | 168 | 175

9. Secondary Outcome: Change From Baseline in Abdominal Pain
Description: Change from baseline in abdominal pain as measured with an 11-point (0-10) Numerical Rating Scale from 0 (No) to 10 (Worst Possible). Baseline is the mean of non-missing abdominal pain scores recorded during the 2-week baseline diary assessment period prior to the first dose of study drug.
Time Frame: Baseline and 12-Week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Matching Placebo | 3.0 mg Plecanatide | 6.0 mg Plecanatide
Number analyzed (Participants) | 354 | 351 | 349
score on a scale
  Baseline | 6.10 (1.793) | 5.94 (1.704) | 5.95 (1.760)
  Week 12 change from baseline | -1.79 (2.196) | -2.11 (2.215) | -2.46 (2.370)

ADVERSE EVENTS:
Description: A total of 1054 patients were randomized, of which two patients did not receive the study drug (6 mg) and resulted in a total of 1052 patients in the Safety population.
Arm/Group | Matching Placebo | 3.0 mg Plecanatide | 6.0 mg Plecanatide
All-Cause Mortality (participants affected / at risk) | 0/354 | 0/351 | 2/347
Serious Adverse Events (participants affected / at risk) | 5/354 | 4/351 | 2/347
Other Adverse Events (participants affected / at risk) | 16/354 | 37/351 | 28/347
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matching Placebo (N=354) | 3.0 mg Plecanatide (N=351) | 6.0 mg Plecanatide (N=347)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increase (Investigations) | 1 (1) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Biplar I disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Drowning (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matching Placebo (N=354) | 3.0 mg Plecanatide (N=351) | 6.0 mg Plecanatide (N=347)
Nasopharyngitis (Infections and infestations) | 7 (7) | 7 (7) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (4) | 4 (4) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 19 (20) | 15 (16)
Nausea (Gastrointestinal disorders) | 3 (3) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes